CLINICAL TRIAL: NCT06170190
Title: A Multicentre, Open-label, Phase 1/2 Study of IBI133 in Subjects With Unresectable, Locally Advanced or Metastatic Solid Tumours
Brief Title: A Multicentre,Study of IBI133 in Subjects WithUnresectable, Locally Advanced or Metastatic SolidTumours
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI133A101
Record Dates: First submitted 2023-11-27; First posted 2023-12-14 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced Unresectable or Metastatic Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open-label：IBI133 monotherapy (Experimental)
  Interventions: Biological: IBI133

INTERVENTIONS:
Biological: IBI133 — IBI133:
  The provisional dose levels are planned to be evaluated, but it is possible for additional and/or intermediate dose levels to be added during the course of the study. Q3W

SUMMARY:
This is a multicentre, open-label, first-in-human, phase 1/2 study of IBI133 in subjects with unresectable, locally advanced or metastatic solid tumours. Phase 1 section includes three parts, IBI133 dose escalation part, and IBI133 monotherapy dose expansion part. The objective of phase 1 section is to identify MTD/recommended dose for expansion (RDE) of IBI133 monotherapy . The objective of phase 2 section is to further explore efficacy, safety and tolerability of IBI133 monotherapy at RDE in specified tumour population. The treatment cycle of the study is defined as every 3 weeks (21 days).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with the ability to understand and give written informed consent for participation in this trial, including all evaluations and procedures as specified by this protocol;
2. Male or female subjects ≥ 18 years old;
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1;
4. Anticipated life expectancy of ≥ 12 weeks;
5. Adequate bone marrow and organ function.
6. Has a documented (histologically- or cytologically-proven), unresectable, locally advanced or metastatic solid tumour that is refractory to or intolerable with standard treatment, or for which no standard treatment is available;

Exclusion Criteria:

1. Participate in any other interventional clinical research except observational (non-interventional) study or in the follow-up phase of the interventional study;
2. Prior HER3 targeted treatment, including but not limited to monoclonal antibody, bispecific antibody, T cell engager, and antibody-drug conjugate.
3. Prior treatment with an antibody-drug conjugate (ADC) which consists of an exatecan derivative that is a topoisomerase I inhibitor (e.g. DS-8201).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) | 21 days after the first dose of IBI133
  DLTs are assessed during the DLT observation period to determine maximum tolerated dose (MTD)and /or recommended phase 2 dose (RP2D)
Safety: Adverse events (AEs);treatment emergent adverse event(TEAEs),serious adverse events(SAEs) | Up to 90 days after the last administration
  Adverse events will be assessed by investigator(s)according to NCI-CTCAE v5.0

SECONDARY OUTCOMES:
maximum concentration (Cmax) | Up to 2 years
  PK parameters maximum concentration(Cmax)of IBI133,total antibody,can will be determined
area under the curve (AUC) | Up to 2 years
  PK parameters clearance rate of IBI133,total antibody,exate can will be determined
clearance rate(CL) | Up to 2 years
  PK parameters clearance rateof IBI133,total antibody,exate can will be determined
half-life (T1/2) | Up to 2 years
  PK parameters half-life of IBI133,total antibody,exate can will be determined
anti-drug antibody (ADA) | Up to 2 years
  the incidence and characterization of ADA OF IBI133 will be determined
Preliminary efficacy including objective response rate (ORR) | Through study completion,Up to 2 years
  ORR is defined as the proportion of subjects with a CR or PR. Number and percentage of subjects with CR or PR will be summarized.
duration of response (DoR) | Through study completion,Up to 2 years
  DoR is defined as the time from the date first achieved CR or PR until the date of first documents disease progression based on RECIST v1.1 or death
disease control rate (DCR) | Through study completion,Up to 2 years
  DCR is defined as the proportion of subjects with a CR, PR or SD, and will be analysed in the same fashion as ORR.
,time to response (TTR) | Through study completion,Up to 2 years
  TTR is defined as the time from the date of first study drug to the date first achieved CR or PR based on RECIST v1.1.
progression free survival (PFS) | Through study completion,Up to 2 years
  PFS is defined as the time from the date of first study drug to death or disease progression based on RECIST v1.1, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool Hospital, Liverpool, New South Wales, Australia